CLINICAL TRIAL: NCT07197918
Title: Prospective Identification of Hypoxic Ischemic Brain Injury Using Portable Magnetic Resonance Imaging
Brief Title: Identification of Brain Injury Using Portable MRI
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000040339; 1R21NS145048-01 (NIH)
Record Dates: First submitted 2025-09-26; First posted 2025-09-30 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrest (CA); Hypoxic-Ischemic Brain Injury
MeSH Terms: conditions — Heart Arrest; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Cardiac arrest with Return of Spontaneous Circulation (ROSC): All enrolled patients will have two to three portable MRIs ( <6 hours, 6-24 hours and one within 12 (+/- 12) hours of conventional MRI) and one conventional MRI. Standard of care will occur per the clinical team and this study will not interfere with standard of care.
  Interventions: Device: portable MRI scanner

INTERVENTIONS:
Device: portable MRI scanner — Participants will receive 2-3 portable MRI scans: <6 hours, 6-24 hours, and within 12 (+/- 12) hours of conventional MRI

SUMMARY:
The goal of this study is to look for brain injury in patients who had a cardiac arrest, using portable brain imaging. The portable nature of this test will also allow for serial imaging so the investigators can understand how brain injury changes over days. The results of this study may allow for bedside imaging to be available at centers without specialized imaging centers and may identify markers of brain injury that help to select the patients most likely to benefit for clinical trials.

DETAILED DESCRIPTION:
Cardiac arrest occurs when the heart stops beating. This can occur for many reasons ranging from a heart attack to a drug overdose. It claims close to 500,000 lives a year. Even though the heartbeat is restored, blood flow to the brain remains below what is required for normal function. Brain injury is common in patients who had a cardiac arrest and few return to independence. Most patients are in a coma following cardiac arrest. Some patients wake up within the first days to week, but most do not. Physicians rely on tests, such as brain imaging, brain wave tests, and lab tests to help predict recovery. Magnetic resonance imaging is a type of brain test used to look for injury to the brain. This type of imaging is not available in community centers and requires transport out of the intensive care unit. Transport can be dangerous in patients who are on life support. New tools have been developed that allow for imaging at the bedside.

These portable machines allow patients to stay connected to all necessary monitoring and decrease interruptions in treatment.

Primary Objective:

A. To evaluate inter-rater agreement of low-field portable MRI as compared to high-field conventional MRI for measuring hypoxic ischemic brain injury severity, using a qualitative MRI scoring system.

B. To acquire early low-field portable MRI (<6 and <24 hours from cardiac arrest) to establish the specificity and positive predictive value of early DWI lesions for predicting hypoxic ischemic brain injury on later conventional MRI.

Secondary Objectives (if applicable):

i. To characterize changes in the regions affected and severity of hypoxic ischemic brain injury on MRI over time.

ii. To identify the impact of early DWI lesions on neurologic prognosis iii. To quantify the incidence of early DWI lesions in post-cardiac arrest patients iv. To describe the feasibility of serial portable MRI in post-cardiac arrest patients

ELIGIBILITY:
Inclusion Criteria:

* Unresponsive immediately after ROSC from IHCA or OHCA
* Age ≥ 18 years of age
* Conventional MRI is clinically indicated
* Treatment with temperature control

Exclusion Criteria:

* MRI contraindication according to the American Heart Association guidelines
* Inability to tolerate supine positioning for 30 minutes
* Diffuse loss of grey-white differentiation and sulcal effacement on head computed tomography within 6 hours of ROSC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comatose adult survivors of out-of-hospital cardiac arrest, treated with temperature control will be enrolled in the emergency department or intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Cortex- DGN HIBI score | up to 6 hours post cardiac arrest, up to 24 hours post cardiac arrest and within 12 (+/- 12) hours of conventional MRI
  Hypoxic ischemic brain injury will be assessed using the Cortex- DGN HIBI score on a scale of 0-40. Higher scores indicate greater injury.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Beekman, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will produce a prospective clinical database and an MRI repository, including serial low-field MRI and a single conventional standard of care MRI. De-identified data will be made available for submission to the NINDS data repository or elsewhere as arranged with the Institute. Data will also be submitted to OpenNeuro
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The scientific data from this study will be shared as soon as possible and no later than the time of an associated publication or the end of the performance period, whichever comes first. Once submitted to the repository, OpenNeuro will manage its availability for an indefinite period of time.
Access Criteria: Requests to access the shared data after the trial is completed will be handled by the NINDS data repository.